CLINICAL TRIAL: NCT00314093
Title: Phase II Evaluation of RFT5-dgA in Patients With Metastatic Melanoma
Brief Title: RFT-5-dgA in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 060137; 06-C-0137; NCT00331461 (obsolete NCT alias)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Melanoma
Keywords: Clinical Response; Stage IV Melanoma; Immunotoxin; T Regulatory Cells; CD25+ Cells; Metastatic Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Drug: RFT5pdgA

SUMMARY:
Background:

* CD4+ cells are white blood cells that regulate the immune system by controlling the strength and quality of the immune response.
* CD25+ cells are a subset of CD4+ cells that suppress or prevent immune responses.
* RFT-5-dgA is an immunotoxin (substance that kills specific cells in the immune system) that kills CD25+ cells.
* In mouse studies, RFT-5-dgA showed anti-tumor activity in animals studies.

Objective: To determine whether the immune system of patients with metastatic melanoma (melanoma that has spread beyond the original site) can cause tumors to shrink if the patients are given RFT-5-dgA to remove their CD25+ cells.

Eligibility: Patients 18 years of age and older with metastatic melanoma whose disease has progressed after receiving standard treatment.

Design:

* Patients receive RFT-5-dgA through a vein every other day for a total of 3 doses (one treatment course). Patients have routine blood tests during the week of treatment.
* Four to 5 weeks after the last dose, patients are evaluated with a physical examination, blood tests and scans and x-rays to evaluate their tumor.
* Patients whose tumor has shrunk or remained stable may be offered additional treatment with RFT-5-dgA up to a total of four courses.
* Patients undergo leukapheresis or have several tubes of blood drawn from a vein to determine the effects of RFT-5-dgA on the immune system. This is done before the first dose of RFT-5-dgA, after the first three doses, and possibly during subsequent treatment courses in those patients who receive additional treatment. For leukapheresis, blood is collected through a needle in an arm vein and flows through a catheter into a machine that separates it into its components by spinning. The white cells are extracted and the rest of the blood is returned through another needle in the other arm.

DETAILED DESCRIPTION:
Background:

* RFT5-dgA is an immunotoxin comprised of the IL-2Ra-specific murine IgG1 antibody RFT5 linked to deglycosylated ricin A chain (dgA) via the sterically hindered heterobifunctional disulfide linker SMPT (4-succinimidyl-oxycarbonyl-a-methyl-a-(2-pyridyldithio)-toluene).
* RFT5-dgA is a recombinant immunotoxin that selectively targets CD25 expressing cells in vivo. Further, treatment of human PBMC with RFT5-dgA in vitro results in the preferential depletion of CD25+ Treg cells.
* Depletion of Treg cells can enhance tumor protection to tumor-associated antigens expressed as self antigens and the RFT5-dgA immunotoxin had potent antitumor effects in SCID mice xenografted with L540 cells which express CD25.
* The MTD established in the phase I trial of RFT5-dgA was 15mg/m(2)/course IV.

Objectives:

* The primary objective is to determine whether objective clinical responses can be obtained in patients with metastatic melanoma following administration of RFT5-dgA.
* Secondary objectives will determine whether changes occur in levels of CD4+CD25+ regulatory T cells (Treg cells) in peripheral blood from before to after treatment and evaluate the toxicity profile of patients treated on this trial.

Eligibility:

* Patients greater than 18 years of age with measurable metastatic melanoma, an expected survival greater than three months, who have progressed after receiving standard therapy will be included.
* Standard clinical laboratory values must be normal for study inclusion and patients may not be pregnant, breast-feeding or require anticoagulation.
* Patients must be willing to undergo leukapheresis.
* Patients with active infections, other major medical disorders, HAMA levels greater than 1 ug/mL, or who have had prior radiotherapy or who have extensive lung disease will be excluded.

Design:

* Patients will receive 3 mg/m(2) RFT5-dgA intravenously every other day for a total of 3 doses (one course).
* Four to five weeks after the last dose, patients will undergo tumor evaluation, evaluation of changes in T-regulatory cells (CD4+CD25+cells and Foxp3 expression), and toxicity assessment.
* One additional course may be administered to patients with stable disease or partial or complete response.
* Up to 41 evaluable patients may be accrued to determine whether theRFT5-dgA can produce a modest response rate targeted to be 20 percent (p1=0.20)
* Enrollment reflects the anticipated enrollment. Actual enrollment is unknown due to no longer having access to the data as records were destroyed

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients age greater than 18 with measurable metastatic melanoma that have an expected survival of greater than three months will be considered. Patients with resectable local/regional disease would undergo standard treatment with surgical resection and will not be eligible.
  2. Patients must be able to understand and give informed consent.
  3. Patients must have progressed while receiving standard therapy which may include IL-2; however, prior IL-2 therapy is not a requirement for enrollment.
  4. Serum creatinine of 1.6 mg/dl or less.
  5. Total bilirubin 2.0 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  6. WBC 3000/mm(3) or greater.
  7. Platelet count 90,000 mm(3) or greater
  8. Serum albumin greater than 2.5 g/dl,
  9. Serum AST/ALT less then 2.5 times normal,
  10. ECOG performance status of 0 or 1 or 2.
  11. For patients greater than 50 years of age or who have a history of cardiovascular disease a thallium stress test is required with EF greater than or equal to 45%.
  12. Patients of both genders must be willing to practice effective birth control during this trial.
  13. Patients must be willing to undergo leukapheresis.

EXCLUSION CRITERIA:

Patients will be excluded:

1. who are undergoing or have undergone in the past 3 weeks any other systemic form of therapy for their cancer.
2. who received RFT5-dgA on another trial.
3. who have uncontrolled concurrent illness including, but not limited to: ongoing or active infection; ongoing or active cardiac disease, such as symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements.
4. who require systemic steroid therapy upon entry into the trial.
5. who are pregnant or breast-feeding.
6. who are known to be positive for hepatitis B(s)AG, hepatitis C or HIV antibody (because of possible immune effects of these conditions).
7. who require chronic anticoagulation.
8. who are 50 years old or greater who do not have a normal stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) with a LVEF less than 45%.
9. who have history of EKG abnormalities, symptoms of cardiac ischemia or arrhythmias who do not have a normal stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) with a LVEF lea than 45%.
10. who have any autoimmune diseases or immunodeficiency (including HIV),or other concurrent malignancies.
11. Who have HAMA levels greater than 1 ug/mL.
12. Who have had prior radiotherapy including radiotherapy to the lung, except for patients who have undergone localized soft tissue radiotherapy.
13. Who have extensive lung disease where greater than 15% of the lung is involved based on CT evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Phan GQ, Yang JC, Sherry RM, Hwu P, Topalian SL, Schwartzentruber DJ, Restifo NP, Haworth LR, Seipp CA, Freezer LJ, Morton KE, Mavroukakis SA, Duray PH, Steinberg SM, Allison JP, Davis TA, Rosenberg SA. Cancer regression and autoimmunity induced by cytotoxic T lymphocyte-associated antigen 4 blockade in patients with metastatic melanoma. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8372-7. doi: 10.1073/pnas.1533209100. Epub 2003 Jun 25. PMID 12826605
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2006-C-0137.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment reflects the anticipated enrollment. Actual enrollment is unknown due to no longer having access to the data as records were destroyed.
Groups:
- No Study Data Available: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed. No study data are available
Period: Overall Study
Arm/Group | No Study Data Available
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed.
Groups:
- Data Not Able to be Obtained: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed
Arm/Group | Data Not Able to be Obtained
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Clinical Responses Can be Obtained in Following Administration of RFT5-dgA
Description: The primary objective is to determine whether objective clinical responses can be obtained in patients with metastatic melanoma following administration of RFT5-dgA
Time Frame: up to one year
Population: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed
Arm/Group | Data Not Able to be Obtained
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine Whether Changes Occur in Levels of CD4+CD25+ Regulatory T Cells (Treg Cells) in Peripheral Blood
Description: Secondary objectives will determine whether changes occur in levels of CD4+CD25+ regulatory T cells (Treg cells) in peripheral blood from before to after treatment and evaluate the toxicity profile of patients treated on this trial.
Time Frame: Before to after treatment
Population: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed
Arm/Group | Data Not Able to be Obtained
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity Profile
Description: as for outcome 2
Population: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed
Arm/Group | Data Not Able to be Obtained
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed
Arm/Group | Data Not Able to be Obtained
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Data Not Able to be Obtained (N=0)
No Data Available (Investigations) | 0 (0) — Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Data Not Able to be Obtained (N=0)
No Data Available (Investigations) | 0 (0) — Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed

LIMITATIONS AND CAVEATS:
Sincere efforts were made to obtain the study data, but were unsuccessful as all study records have been destroyed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes